CLINICAL TRIAL: NCT06823674
Title: The Relationship of Core Endurance With Cervical Stabilization and Proprioception in Women With and Without Pilates Exercise
Status: Active, not recruiting | Type: Observational
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Selin Kalın, Physiotherapist Selin Kalın, Istanbul Arel University
Other Study IDs: E-52857131-050.04-591162
Record Dates: First submitted 2025-01-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pilates Exercise
Keywords: core endurance, pilates, stabilization, proprioception

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tests were performed to measure core endurance, cervical stabilization and cervical proprioception. No specimen samples were collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women Who Don't Do Pilates: 20 women aged 20-50 years who were sedentary according to the International Physical Activity Questionnaire and had not participated in any pilates or yoga exercise group in the last 1 year
  Interventions: Other: core endurance test; Other: cervical stabilization test; Other: cervical proprioception test
- Women Doing Pilates: 20 female volunteers between the ages of 20-50, practicing Pilates at least 2 days a week for at least 12 weeks
  Interventions: Other: core endurance test; Other: cervical stabilization test; Other: cervical proprioception test

INTERVENTIONS:
Other: core endurance test — The study group was selected from women who did pilates exercises 2 days a week for at least 12 weeks under the supervision of a physiotherapist, while the control group was selected from women who did not participate in any pilates, yoga or exercise program in the last 1 year and were sedentary according to the International Physical Activity Questionnaire. Lateral Bridge Test, Static Trunk Extension Test, Trunk Flexors Endurance Test, Cervical Joint Position Error Test, Cervical Region Deep Flexor Muscle Endurance Tests were applied to the participants and Craniocervical Flexion data of the participants were evaluated with Stabilizer Pressure Biofeedback Device.
Other: cervical stabilization test — The study group was selected from women who did pilates exercises 2 days a week for at least 12 weeks under the supervision of a physiotherapist, while the control group was selected from women who did not participate in any pilates, yoga or exercise program in the last 1 year and were sedentary according to the International Physical Activity Questionnaire. Lateral Bridge Test, Static Trunk Extension Test, Trunk Flexors Endurance Test, Cervical Joint Position Error Test, Cervical Region Deep Flexor Muscle Endurance Tests were applied to the participants and Craniocervical Flexion data of the participants were evaluated with Stabilizer Pressure Biofeedback Device.
Other: cervical proprioception test — The study group was selected from women who did pilates exercises 2 days a week for at least 12 weeks under the supervision of a physiotherapist, while the control group was selected from women who did not participate in any pilates, yoga or exercise program in the last 1 year and were sedentary according to the International Physical Activity Questionnaire. Lateral Bridge Test, Static Trunk Extension Test, Trunk Flexors Endurance Test, Cervical Joint Position Error Test, Cervical Region Deep Flexor Muscle Endurance Tests were applied to the participants and Craniocervical Flexion data of the participants were evaluated with Stabilizer Pressure Biofeedback Device.

SUMMARY:
The aim of this study was to investigate the relationship between core endurance and cervical stabilization and proprioception in women with and without Pilates exercise. The study was conducted with 40 volunteer female participants aged 20-50 years. The study group was selected from women who did Pilates exercises 2 days a week for at least 12 weeks under the supervision of a physiotherapist, while the control group was selected from women who did not participate in any Pilates, yoga or exercise program in the last 1 year and were sedentary according to the International Physical Activity Questionnaire. Lateral Bridge Test, Static Trunk Extension Test, Trunk Flexor Endurance Test, Cervical Joint Position Error Test, Cervical Region Deep Flexor Muscle Endurance Tests were applied to the participants and Craniocervical Flexion data of the participants were evaluated with Stabilizer Pressure Biofeedback Device and the results were recorded. These results indicate that high performance in core endurance is associated with improved performance in cervical stabilization. As a result of this study, it was concluded that Pilates has a significant effect on core endurance, cervical stabilization and proprioception in women.

ELIGIBILITY:
Inclusion Criteria:

* Being between 20-50 years old
* Volunteering to participate in the study
* Having practiced Pilates at least 2 days a week for at least 12 weeks for the study group
* For the control group, not having participated in any pilates, yoga or exercise program in the last year and being sedentary according to the International Physical Activity Questionnaire

Exclusion Criteria:

* Presence of pain during assessments
* Cervical and/or lumbar disc herniation
* Spine pathology

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female participants aged 20-50 years
Study Population: Group of 20 participants doing pilates exercise 20 participants in the group without pilates exercise
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Core Muscle Endurance between Pilates and Non-Pilates Groups Mann Whitney U Test Analysis | 01.05.2024- 20.07.2024
  The endurance of the core muscles was used to assess the static resistance of the core region with three tests evaluating the trunk flexors, trunk extensors and lateral bridge exercise. Lateral Bridge Test, Static Trunk Extension Test (Sorensen Test) and Trunk Flexors Endurance Test were evaluated, measurements were recorded in seconds using a stopwatch. The tests were repeated twice and the best result value was recorded. The test was terminated when the person administered was unable to maintain the position or when the person said that they could not continue the test
Mann Whitney U Test Analysis of Deep Neck Flexor Muscle Endurance Assessment Between Pilates and Non-Pilates Exercise Groups | 01.05.2024- 20.07.2024
  The participant was positioned in the supine hook position with hands relaxed on the abdomen. The participant was instructed to pull his/her chin inwards (chin tuck) and lift his/her head off the bed while maintaining this position (approximately 2.5 cm). The participant was asked to maintain this position for as long as possible without distortion and the time to maintain the position was recorded in seconds. In order to perform the test correctly, the test was demonstrated to the individuals in a practical way before starting the test. The test duration was kept short to prevent pain and fatigue of the participant. The test was stopped when the jaw position (craniocervical flexion movement and jaw) was lost and sudden pain increased and the subject did not want to continue the test. A single test was performed and the time was recorded in seconds.
Chi-Square Test Analysis of Completion Distributions of Stages in Craniocervical Flexion Measurement with Stabilizer Pressure Biofeedback Device According to Groups | 01.05.2024- 20.07.2024
  In our study, after the participants were placed supine on the examination bed, the pressure cell was placed under the nape of the neck without inflation. The cell was inflated to 20 mmHg, taking care not to slide the cell to the lower cervical region. The participant was asked to press the chin towards the neck without lifting the head as if saying 'yes' (posterior cervical tilt). The participant was instructed to place the tongue on the upper palate, bring the lips together but keep the teeth slightly apart.
  The test consists of 5 stages. The value of the stabiliser device, which was set at 20 mmHg, was asked to increase by 2 mmHg at each stage until it reached 30 mmHg (20- 22- 24- 26- 28- 30 mmHg). The participant was asked to stay at each pressure value for 30 s and to complete the test by giving 30 s rest time after each pressure. The test was terminated at the stage where the participant could not complete the pressure value that he/she should keep constant for 30 s.
Cervical Joint Position Error Test (Cervical Proprioception Assessment) Between Pilates and Non-Pilates Exercise Groups | 01.05.2024- 20.07.2024
  It is a measurement tool used to clinically assess participants' cervicocephalic proprioception ability. Cervicocephalic proprioception describes the sense of position of one's head and neck in space. It measures the ability of a blindfolded participant to accurately return the head position to a predetermined neutral point after cervical joint movement

CONTACTS AND LOCATIONS:
Overall Officials: Selin K Kalın, Principal Investigator — İstanbul Arel Üniversitesi
Locations (1):
- Burak Sapmaz Fizyoterapi ve Danışmanlık Merkezi, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Çalışma boyunca toplanan tüm IPDler paylaşılabilir.